CLINICAL TRIAL: NCT02390934
Title: Single Arm Phase II Trial Evaluating the Efficacy of Radium 223 in Radioactive Iodine Refractory Bone Metastases From Differentiated Thyroid Cancer
Brief Title: Efficacy of Radium 223 in Radioactive Iodine Refractory Bone Metastases From Differentiated Thyroid Cancer
Acronym: RAD-THYR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-001070-34; 2014/2110 (Other: CSET number)
Record Dates: First submitted 2014-10-01; First posted 2015-03-18 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Thyroid Cancer
Keywords: Radium 223; bone metastases
MeSH Terms: conditions — Thyroid Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radium 223 (Experimental): Radium-223 (Xofigo®) will be supplied in vials as a ready-to-use solution for intravenous administration. The activity (administered radioactivity) will be 50 kBq/kg b.w., and multiple treatment activities up to 6 injections will be administered at intervals of 4 weeks.
  Interventions: Radiation: Radium 223

INTERVENTIONS:
Radiation: Radium 223
  Other Names: Xofigo

SUMMARY:
The purpose of this Phase II single-arm study is to evaluate the efficacy of Radium-223 in treating bone lesions from differentiated thyroid cancer that are I-131 refractory. Based on the results of the phase III trial, the protocol using an injection of Radium-223 activity of 50 kBq/kg b.w. given 6 times at 4 weeks interval will be applied. The end point of this study will be the evaluation of Radium-223 efficacy one month after 3 administrations, i.e. at 3 months after the first injection. If disease progression at that time is excluded, patients will be treated with 3 further injections for a total of 6 administrations of Radium-223. The principal response criterion at 3 and 6 months will be the metabolic response on FDG PET/CT, but other imaging techniques will also be performed: axial skeleton MRI, 99mTc-HMDP bone scan and FNa PET/CT. Axial skeleton MRI is the reference for soft tissue study. 99mTc- HMDP bone scan is the most used and available routine tool to detect bone metastases in cancer patients, but its sensitivity in patients with bone metastases from thyroid cancer is low, because most lesions are lytic [23]. 18FNa PET/CT shows higher sensitivity than 99mTc-HMDP bone scan to detect bone lesions in cancer patients and is able to detect micrometastases that are not seen on bone scan [24] [25]. Preliminary results show some interest of using this tracer to evaluate the sclerotic component of bone metastases from thyroid cancer [26]. Furthermore preliminary data show that FNa PET/CT can be useful to quantify response to Radium-223 in prostate cancer. In only five patients evaluated by FNa PET/CT at baseline, 6 weeks and 12 weeks after 100 KBq/Kg of Radium-223, semiquantitative analysis by SUV max showed a relationship between PSA and SUV max level decrease in 3 patients (-44%, -31%, -27% vs -52%, -75, and -49% respectively) [27].

Finally bone metastases that are visible on morphological imaging (CT scan or on RI) are frequently submitted to local treatment modalities, and this may induce fibrosis and recalcification. Therefore, already treated metastases and not treated metastases will be studied separately as two separate subgroups of target lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Affiliated to a social security regimen ;
2. Patients with histologically confirmed differentiated thyroid cancer (papillary, follicular including Hurthle cell or poorly differentiated) ;
3. Iodine refractory disease defined by the absence of radioiodine uptake in at least one lesion or progression of the disease within 14 months after a radioactive iodine (RAI) treatment or persistent disease after the administration of a cumulative activity of 22GBq I 131 ;
4. Age ≥18 years ;
5. Eastern Cooperative Oncology Group performance status 0-2 ;
6. Life expectancy longer than 3 months ;
7. Presence of at least one bone metastasis visible on CT scan or axial skeleton (AS) MRI and not requiring urgent locoregional treatment ;
8. Presence of at least one bone metastasis with uptake on FDG PET/CT ;
9. Presence of at least one bone metastasis with increased uptake on 99mTc HMDP bone scintigraphy or FNa PET/CT
10. Low likelihood of an indication for systemic treatment within the next 6 months, as defined by the absence of soft tissue distant metastases or by the presence of only small (<1cm) soft-tissue metastases, or larger (>1 cm) but stable soft tissue metastases within 6 months prior to inclusion in the present protocol ;
11. Adequate haematological (neutrophils ≥1,5×109/L; platelets ≥100×109/ L; haemoglobin > 9g/dL), renal (creatinine <1,5×upper limit of normal range), and hepatic (total bilirubin < 1.5 institutional upper limit of normal), aspartate aminotransferase and alanine aminotransferase <2,5×upper limit of normal range in the absence of liver metastases or <5×upper limit of normal range in case of liver metastases) functions ;
12. Patients receiving bisphosphonates or anti-RANK ligand (Denosumab) are allowed but patients should have received at least 2 administrations prior to Radium-223 administration and these treatments will be continued during Radium-223 treatment ;
13. Blood negative pregnancy test in women of childbearing potential within 30 days prior to treatment initiation. Both men and women (of childbearing potential) who are sexually active must use adequate contraception during and for at least 6 months post-treatment ;
14. Patient who is fully informed, able to comply with the protocol and who signed the informed consent.

Exclusion Criteria:

1. Patients with another malignancy that is not in remission for at least 2 years (except for in situ cervix uterine cancer, basocellular skin cancer) ;
2. Treatment with any investigational drug or with a TKI within the previous 4 weeks, or planned during the treatment period ;
3. Treatment with cytotoxic chemotherapy within the previous 4 weeks, or planned during the treatment period, or failure to recover from adverse events due to cytotoxic chemotherapy administered more than 4 weeks before the study initiation ;
4. Previous systemic therapy with radionuclides, including strontium-89, samarium-153, rhenium-186, rhenium-188 or radium-223 ;
5. Patients with imminent or established spinal cord compression based on clinical findings and/or MRI and/or immediate need for local radiotherapy ;
6. Patients with progressive visceral metastases according to RECIST 1.1 criteria assessed by CT scan and/or symptomatic brain metastases within 6 months prior to study initiation ;
7. Patient already included in other clinical trial ;
8. Pregnant or breast feeding women ;
9. Fecal or urinary unmanageable incontinence ;
10. Bone marrow dysplasia, uncontrolled diabetes or infection, NYHA Class III or IV cardiac disorders, fecal incontinence and symptomatic intestinal disease (such as Crohn disease or ulcerative colitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Metabolic response (PERCIST criteria) | Assessed 1 months after 3 monthly injections of Radium 223
  Metabolic response according to PERCIST criteria in up to five lesions on FDG PET/CT performed 1 month after 3 monthly injections of Radium 223

SECONDARY OUTCOMES:
Pain response (numerical rating scale) | Assessed every 30 days following the first Radium 223 up to 7 months
  evaluated on a 0-to-10 numerical rating scale completed by the patients
Partial pain response (improvement ≥30% and <50% pain score) | Assessed every 30 days following the first Radium 223 up to 7 months
  Partial pain response is defined as an improvement ≥30% and <50% of the worst pain compared to score at baseline. Complete pain response is defined as an improvement ≥50% of the worst pain score compared to score at baseline
ECOG performance status | Assessed every 30 days following the first Radium 223 up to 7 months
Changes in Quality of life (QLQ-C30 and QLQ-BM22 questionnaires) | Assessed every 30 days following the first Radium 223 up to 7 months
  evaluated with the QLQ-C30 and QLQ-BM22 questionnaires
Time to occurrence of first skeletal-related events | Assessed every 30 days following the first Radium 223 up to 7 months
  ) confirmed by imaging defined as: (i) local progression with indication for local treatment such as surgery, thermoablation, cement injection, external beam radiation, or (ii) pathological fracture, spinal cord compression (iii) appearance of new bone lesions.
Overall survival | Assessed every 30 days following the first Radium 223 up to 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie LEBOULLEUX, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Deandreis D, Maillard A, Zerdoud S, Bournaud C, Vija L, Sajous C, Terroir M, Leenhardt L, Schlumberger M, Borget I, Leboulleux S. RADTHYR: an open-label, single-arm, prospective multicenter phase II trial of Radium-223 for the treatment of bone metastases from radioactive iodine refractory differentiated thyroid cancer. Eur J Nucl Med Mol Imaging. 2021 Sep;48(10):3238-3249. doi: 10.1007/s00259-021-05229-y. Epub 2021 Feb 23. PMID 33619600